CLINICAL TRIAL: NCT01978314
Title: A Single-Center Prospective Study Evaluating the FAST Measured Glomerular Filtration Rate (mGFR) Test™ in Adults With Preserved Kidney Function and Impaired Kidney Function With Comparison to Iohexol Clearance Methods
Brief Title: FAST GFR: Pilot Study to Evaluate the Safety of the FAST GFR Test in Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FAST BioMedical (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FAST mGFR -002; 1R44DK093274-01 (NIH)
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Disease; Acute Kidney Injury
Keywords: Chronic Kidney Disease; Acute Kidney Injury; AKI; CKD; Plasma Volume; GFR; Glomerular Filtration Rate; Blood volume; mGFR; measured GFR; kidney biomarker; renal disease; renal biomarker; Renal function; kidney function; organ function; kidney monitor; kidney device
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This pilot study was a prospective, open-label, single site study designed to evaluate the safety of the FAST mGFR Test™ in healthy adult volunteers, patients with varying degrees of renal impairment and hemodynamically stable AKI.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): eGFR renal function ≥60 mL/min for normal function 75 mg / 6mL VFI™ and 5mL of Iohexol
  Interventions: Device: 75 mg / 6 mL VFI™
- Cohort 2 (Experimental): eGFR renal function 30-59 mL/min for stage 3, moderate CKD 75 mg / 6mL VFI™ and 5mL of Iohexol
  Interventions: Device: 75 mg / 6 mL VFI™
- Cohort 3 (Experimental): eGFR renal function 15-29 mL/min for stage 4, severe CKD 75 mg / 6mL VFI™ and 5mL of Iohexol
  Interventions: Device: 75 mg / 6 mL VFI™
- Cohort 4 (Experimental): a diagnosis of either RIFLE stage I or Acute Kidney Injury Network (AKIN) stage 2 AKI 75 mg / 6mL VFI™ and 5mL of Iohexol
  Interventions: Device: 75 mg / 6 mL VFI™
- Cohort 5 (Experimental): eGFR renal function ≥60 mL/min for normal function 75 mg / 6mL VFI™ and 5mL of Iohexol
  Interventions: Device: 75 mg / 6 mL VFI™

INTERVENTIONS:
Device: 75 mg / 6 mL VFI™ — Visible fluorescent injectate, a mixture of two different molecular weight carboxymethyl dextran molecules (5 kD and 150 kD) with different fluorescent dye molecules attached.

SUMMARY:
This is a single site study designed to evaluate the FAST mGFR Test™ in healthy adult volunteers, patients with varying degrees of chronic kidney disease (CKD), and patients with acute kidney injury (AKI).

DETAILED DESCRIPTION:
A rapid and accurate measurement of glomerular filtration rate (GFR) is important in acute kidney injury (AKI) and chronic kidney disease (CKD) for assessment of impairment, diagnosis, and prompt treatment. FAST BioMedical is an emerging technology company whose mission is to quantify clinically meaning ful physiological parameters that have been difficult or impossible to measure. GFR is the most clinically relevant metric for understanding renal function, as it is the rate by which the kidney is able to filter waste products in the bloodstream. The FAST mGFR is for direct measurement of GFR that relies on reading the ratio of fluorescent markers attached to different size dextran molecules introduced into the bloodstream. The test is intended as an adjunct to current methods utilized to assess kidney function.

ELIGIBILITY:
Inclusion Criteria for Groups 1-3:

* Female subjects: women must have a negative urine pregnancy test at screening and before dosing on Visit 2 and be either confirmed by the Investigator to be infertile or using a reliable method of contraception Male subjects: reproductively active men must agree to either practice abstinence or utilize adequate contraception.
* Ages 19 to 75
* Subject's screening must fall into one of the available categories of estimated glomerular filtration rate (eGFR) renal function: ≥ 60 mL/min for stage normal function; 30-59 mL/min for stage 3, moderate CKD; 15-29 mL/min for stage 4, severe CKD,
* Patients must not be on inotropes or vasopressors, and must be absent of significant hemodynamic instabilities.
* Patients must have ceased use of the following:

  * nonsteroidal anti-inflammatory drugs - 6 days prior,
  * herbal supplements - 6 days prior to testing and
  * cimetidine and trimethoprim - 14 days prior to testing.
* Ability to comply with study conditions

Inclusion Criteria for Group 4:

- Female subjects; women must have a negative urine pregnancy test at screening and before dosing on Visit 2 and be either confirmed by the Investigator to be infertile or using a reliable method of contraception.

Male subjects: reproductively active men must agree to either practice abstinence or utilize adequate contraception.

* Ages 19 to 75
* For cohort 4: patients diagnosed with [either RIFLE stage I or Acute Kidney Injury Network (AKIN) stage 2 AKI]
* Patients must not be on inotropes or vasopressors, and must be absent of significant hemodynamic instabilities.
* Patients must be without evidence of clinically significant liver dysfunction
* Ability to comply with study conditions

Exclusion Criteria for Groups 1-3:

* Positive history of any clinically significant allergic or negative reactions, side effects, or anaphylaxis to sulfa, iodine, dyes, shellfish, isotopes or dextran molecules
* Previous history of nephrectomy or kidney transplant
* A body weight below 40kg
* A body mass index <17 or >40
* Subjects using Coumadin (Warfarin) who have an INR >4 at Screening or pre-dose on Visit 2
* Past history of liver disease or screening Liver Function tests which exceed 1.5 times the upper limit of normal or an albumin of < 2mg/dl.
* Clinically significant illness within 4 weeks or a clinically significant infection within 4 weeks of screening
* Received blood, donated blood, have clinically significant on-going bleeding, changing haemoglobin, or experienced significant blood loss within 2 weeks of dosing
* Subjects with significant abnormal findings upon physical examination, vital signs, ECG, or clinical laboratory results at Screening
* Subjects with a supine blood pressure after resting for at least 5 minutes outside the 90-145 (systolic) or mmHg or 50-95 mmHg (diastolic) range
* Subjects with a supine (ECG) heart rate outside 45-105 beats/min after resting for at least 5 minutes.
* Subjects with a known or suspected history of drug or alcohol misuse within 6 months prior to screening, subjects who have consumed alcohol within 48 hours of dosing, or subjects who the Investigator believes to be unfit to participate in the study due to abuse of illegal or controlled substances.
* Subjects who had a positive result for Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCVAb) screen.
* Subjects who have been diagnosed with acquired immune deficiency syndrome (AIDS), or test positive for human immunodeficiency virus (HIV).
* Subjects who participated in another clinical trial less than 1 month prior to dosing, or who are currently enrolled in another clinical trial.
* Subjects who have any condition that:

  * Would make him/her, in the opinion of the Investigator, unsuitable for the study
  * Whose condition is likely to deteriorate
  * Who, in the opinion of the Investigator, is not likely to complete the study for any reason

Exclusion Criteria for Group 4:

* Positive history of any clinically significant allergic or negative reactions, side effects, or anaphylaxis to sulfa, iodine, dyes, shellfish, isotopes or dextran molecules
* Previous history of nephrectomy or kidney transplant
* A body weight below 40kg
* A body mass index <17 or >40
* Current use of prescribed anticoagulants
* Past history of liver disease or screening Liver Function tests which exceed 1.5 times the upper limit of normal or an albumin of < 2mg/dl.
* Received blood, donated blood, have clinically significant on-going bleeding, changing haemoglobin, or experienced significant blood loss within 2 weeks of dosing
* Subjects with a supine blood pressure after resting for at least 5 minutes outside the 90-145 (systolic) or mmHg or 50-95 mmHg (diastolic) range
* Subjects with a supine (ECG) heart rate outside 45-105 beats/min after resting for at least 5 minutes.
* Subjects with a known or suspected history of drug or alcohol abuse within 6 months prior to admission, who have a positive drug test or alcohol test, or who have consumed alcohol within 24 of testing
* Subjects who had a positive result for Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCVAb) screen.
* Subjects who have been diagnosed with acquired immune deficiency syndrome (AIDS), or test positive for human immunodeficiency virus (HIV).
* Subjects who participated in another clinical trial less than 1 month prior to dosing, or who are currently enrolled in another clinical trial.
* Subjects who have any condition that:

  * Would make him/her, in the opinion of the Investigator, unsuitable for the study
  * Whose condition is likely to deteriorate
  * Who, in the opinion of the Investigator, is not likely to complete the study for any reason

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana V Rizk, M.D, Principal Investigator — University of Alabama Birmingham, 205-934-9509, drizk@uab.edu
Locations (1):
- University of Alabama Birmingham, Division of Nephrology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang E, Meier DJ, Sandoval RM, Von Hendy-Willson VE, Pressler BM, Bunch RM, Alloosh M, Sturek MS, Schwartz GJ, Molitoris BA. A portable fiberoptic ratiometric fluorescence analyzer provides rapid point-of-care determination of glomerular filtration rate in large animals. Kidney Int. 2012 Jan;81(1):112-7. doi: 10.1038/ki.2011.294. Epub 2011 Aug 31. PMID 21881552

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1; Cohort 5: eGFR renal function ≥60 mL/min for normal function
- Cohort 2: eGFR renal function 30-59 mL/min for stage 3, moderate CKD
- Cohort 3: eGFR renal function 15-29 mL/min for stage 4, severe CKD
- Cohort 4: a diagnosis of either RIFLE stage I or Acute Kidney Injury Network (AKIN) stage 2 AKI
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 8 | 8 | 8 | 1 | 8
Completed | 8 | 8 | 8 | 1 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1; Cohort 5: Estimated GFR (mL/min)
  ≥60 mL/min/1.73m2 BSA
- Cohort 2: Estimated GFR (mL/min) 30-59 mL/min/1.73m2 BSA
- Cohort 3: Estimated GFR (mL/min) 15-29 mL/min/1.73m2 BSA
- Cohort 4: Estimated GFR (mL/min) sCr: ≥2-fold increase or eGFR: >50% decrease compared to baseline
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 8 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 1 | 8 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (5.19) | 56.6 (7.03) | 55.6 (17.74) | 63.0 (0) | 31.8 (14.10) | 46.98 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 0 | 8
  Male | 5 | 6 | 6 | 0 | 8 | 25
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 1 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product or investigational medical device.
Time Frame: Baseline through day 22
Population: Intent-to-treat subject population
Measure: Number; unit: participants
Groups:
- Cohort 4: sCr: ≥2-fold increase or eGFR: >50% decrease compared to baseline
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 8
participants | 3 | 4 | 6 | 1 | 5

2. Primary Outcome: Number of Adverse Events Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: as for outcome 1
Time Frame: Baseline through day 22
Population: Intent-to-treat subject population
Measure: Number; unit: adverse events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 8
adverse events
  Number of treatment-emergent adverse events | 5 | 6 | 9 | 3 | 14
  Number of serious treatment-emergent adverse event | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Cmax of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: Cmax = maximum observed concentration occurring at Tmax
Time Frame: PK parameters were evaluated using samples collected pre and post dose at day 2, as well as post dose on days 4, 8, 15, 22.
Population: Intent-to-treat subject population analyzed. PK was not evaluated in Cohort 1 due to a contamination problem caused by the sample collection catheter used in this cohort. In addition, PK data was not collected for the single subject dosed in Group 4.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
ng/mL
  FD001 |  | 8949 (1350) | 9725 (1847) |  | 9336 (1553)
  FD003 |  | 9569 (1809) | 10906 (2307) |  | 12663 (2680)

4. Secondary Outcome: Tmax of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: Tmax = time of maximum observed concentration
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
hr
  FD001 |  | 0.281 (0.0884) | 0.273 (0.0947) |  | 0.25 (0)
  FD003 |  | 4.33 (8.16) | 0.335 (0.27) |  | 2.64 (3.16)

5. Secondary Outcome: AUClast of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: AUClast = area under the concentration-time curve (time 0 to last sample with a quantifiable measurable concentration)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng∙hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
ng∙hr/mL
  FD001 |  | 37594 (12938) | 74317 (27069) |  | 18681 (2066)
  FD003 |  | 1701850 (276886) | 1642731 (443350) |  | 1710348 (355518)

6. Secondary Outcome: AUCall of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: AUCall = area under the concentration-time curve (time 0 to last scheduled sample)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng∙hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
ng∙hr/mL
  FD001 |  | 42462 (12128) | 80058 (25030) |  | 19924 (2441)
  FD003 |  | 1701850 (276886) | 1642731 (443350) |  | 1710348 (355518)

7. Secondary Outcome: AUCinf of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: AUCinf = area under the concentration-time curve (time 0 extrapolated to infinity based on the last observed concentration)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng∙hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
ng∙hr/mL
  FD001 |  | 38844 (12960) | 76554 (26430) |  | 19127 (2107)
  FD003 |  | 1821296 (302728) | 1756948 (503557) |  | 1755162 (366071)

8. Secondary Outcome: T1/2, z of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: T1/2 = terminal half-life = ln(2)/λz
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
hr
  FD001 |  | 9.48 (4.28) | 18.3 (12.6) |  | 5.64 (1.23)
  FD003 |  | 123 (38.9) | 125 (32.8) |  | 90.9 (10.4)

9. Secondary Outcome: Vz of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: Vz = volume of distribution based upon terminal phase
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
mL/m^2
  FD001 |  | 8343 (1733) | 7907 (2613) |  | 11451 (3430)
  FD003 |  | 1177 (293) | 1384 (644) |  | 1018 (208)

10. Secondary Outcome: Vss of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: Vss = volume of distribution at steady state
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
mL/m^2
  FD001 |  | 5430 (781) | 5464 (1425) |  | 6599 (4289)
  FD003 |  | 1039 (299) | 1132 (274) |  | 937 (181)

11. Secondary Outcome: CL of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: CL = total body clearance
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr/m^2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
mL/hr/m^2
  FD001 |  | 677 (190) | 143 (39.5) |  | 1404 (242)
  FD003 |  | 6.82 (1.26) | 7.65 (2.67) |  | 7.74 (1.14)

12. Secondary Outcome: Cmax/Dose of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: Cmax/Dose = maximum observed concentration occurring at Tmax/Dose
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: [(ng/mL)/(mg/m^2)]
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
[(ng/mL)/(mg/m^2)]
  FD001 |  | 369 (43.1) | 73.8 (18.7) |  | 354 (55)
  FD003 |  | 787 (125) | 877 (135) |  | 956 (197)

13. Secondary Outcome: AUCinf/Dose of FD001 and FD003 Following Administration of VFI™ in Patients With Varying Degrees of Kidney Function
Description: AUCinf/Dose = area under the concentration-time curve (time 0 extrapolated to infinity based on the last observed concentration)/Dose
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: [(ng∙hr/mL)/(mg/m^2)]
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 8 | 8 | 0 | 8
[(ng∙hr/mL)/(mg/m^2)]
  FD001 |  | 1641 (590) | 1071 (34.6) |  | 731 (129)
  FD003 |  | 150220 (22006) | 141337 (35933) |  | 131599 (19656)

14. Secondary Outcome: To Compare the Results From the GFR Determined From the FAST VFI™ to GFR Derived From Iohexol Clearance Methods.
Description: This analysis will compare estimates of kidney function derived from the results of FAST VFI™ to those derived through conventional Iohexol clearance methods.
Time Frame: Baseline through Day 22
Population: The subject in Cohort 4 did not receive Iohexol. One subject in Cohort 5 withdrew from the study before receiving Iohexol. Samples were missing for 1 subject in each of Cohorts 1 and 3.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 8
mL/min
  VFI mGFR | 83.20 (16.967) | 42.89 (5.810) | 30.17 (5.174) | 70.86 (0) | 65.17 (10.065)
  Iohexol GFR: number analyzed (Participants) | 7 | 8 | 7 | 0 | 7
  Iohexol GFR | 119.25 (9.898) | 57.52 (15.816) | 31.76 (8.340) |  | 110.52 (12.675)

15. Secondary Outcome: To Evaluate the Correlation Between FAST's Plasma Volume Method and Standard Clinical Estimates of Plasma Volume.
Description: This analysis will compare estimates of plasma volume derived by FAST's plasma volume method with that derived using the conventional Nadler's Formula for plasma volume.
Time Frame: Baseline through day 22
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 8
mL
  FAST Plasma Volume | 3251.088 (452.6180) | 2926.941 (568.1260) | 2816.244 (533.7910) | 6046.770 (0) | 2415.950 (569.1105)
  Nadler's Formula Plasma Volume | 2859.671 (313.2253) | 3103.431 (443.1221) | 3150.045 (393.3610) | 5297.820 (0) | 2805.234 (412.2505)

ADVERSE EVENTS:
Time Frame: Baseline through day 22.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/1 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/1 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 4/8 | 6/8 | 1/1 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=8) | Cohort 3 (N=8) | Cohort 4 (N=1) | Cohort 5 (N=8)
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctival Oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Miosis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 2 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Potassium Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac Murmur (Investigations) | 0 | 1 | 0 | 0 | 0
Liver Palpable Subcostal (Investigations) | 0 | 0 | 0 | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Too restrictive entry criteria for enrollment into the AKI cohort and the expiry of the clinical VFI led to a decision, in consultation with FDA, to stop the study prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less